CLINICAL TRIAL: NCT07144189
Title: Artificial Intelligence-Based Assessment of Low-Gradient Aortic Stenosis Severity Using Echocardiographic Images
Brief Title: AI Assessment of Low-Gradient Aortic Stenosis Severity Based on Echocardiography
Acronym: ASAI-POL
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: The Institute of Bioorganic Chemistry, Polish Academy of Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4.35/VI/25
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: Low-gradient Aortic Stenosis; Aortic Stenosis
Keywords: low-gradient aortic stenosis; Echocardiography; Artificial intelligence; Cardiac imaging; Machine learning
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with suspected significant low-gradient aortic stenosis.: Approximately 300 patients with suspected significant low-gradient aortic stenosis undergoing standard echocardiographic evaluation between 2025 and 2026. Echocardiographic images will be secondarily analyzed by the AI model to classify stenosis as severe or moderate. The AI results will be compared with physicians assessments. No intervention or modification of clinical care is involved.
  Interventions: Diagnostic Test: AI diagnostic test for severe low-gradient aortic stenosis

INTERVENTIONS:
Diagnostic Test: AI diagnostic test for severe low-gradient aortic stenosis — All participants will undergo standard transthoracic echocardiography performed for clinical indications. Echocardiographic images will be analyzed both by experienced physicians and by the investigational AI model. Additional diagnostic tests (such as cardiac CT, low-dose dobutamine stress echocardiography or transesophageal echocardiography) may be performed if clinically indicated, according to current guideline recommendations. The AI-derived results will not influence clinical decision-making.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an artificial intelligence (AI) model developed by the investigators for identifying severe low-gradient aortic valve stenosis. Accurate assessment of stenosis severity is crucial for proper qualification for surgical treatment. It is expected that the use of AI will improve diagnostic accuracy and thereby support better clinical outcomes.

Patients with suspected significant low-gradient aortic stenosis will be enrolled. The study is observational and involves no additional risk for participants. Standard imaging studies performed for clinical indications will be additionally analyzed by the AI model, which will classify aortic stenosis as severe or moderate. The model's results will not influence the clinical management of participants but will be compared with physicians' assessments to validate its diagnostic performance.

The study will be conducted in 2025-2026. The findings will provide insights into the usefulness of AI in the diagnosis of severe aortic stenosis and may contribute to the development of advanced clinical decision-support tools.

DETAILED DESCRIPTION:
This study is a prospective multicenter observational validation of an artificial intelligence (AI) model for differentiating severe low-gradient from moderate aortic stenosis using transthoracic echocardiography images. The model, developed and published by the investigators, demonstrated promising diagnostic performance in retrospective data. In the present trial, approximately 300 participants with suspected significant low-gradient aortic stenosis will be enrolled during 2025-2026. Standard imaging studies performed for clinical indications will be analyzed by the AI model, which will classify aortic stenosis as severe or moderate. The AI-derived results will not influence clinical decision-making but will be compared with physicians assessments to evaluate diagnostic accuracy and reproducibility in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical suspicion of significant low-gradient aortic stenosis
* Echocardiographic examination performed for clinical indications
* Ability to provide informed consent

Exclusion Criteria:

* Previous aortic valve intervention (surgical or transcatheter)
* Inadequate image quality precluding echocardiographic analysis
* Concomitant severe valvular disease (severe mitral stenosis or mitral/aortic regurgitation) that could confound assessment
* Patients unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients (≥18 years) diagnosed in the Echocardiography Laboratory of the National Institute of Cardiology in Warsaw, Department of Valvular Heart Disease. Eligible participants will be those referred for echocardiographic evaluation due to clinical suspicion of significant low-gradient aortic stenosis. Standard-of-care imaging performed for clinical indications will be analyzed. Approximately 300 patients are expected to be enrolled between 2025 and 2026. Patients with previous aortic valve intervention (surgical or transcatheter) or other exclusion criteria will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) describing the sensitivity-specificity relationship of the AI model. | At the time of the nearest Heart Team meeting following the echocardiographic examination (typically within 1 week).
  AUC will be calculated to assess the ability of the AI model to differentiate between severe low-gradient and moderate aortic stenosis. The analysis will use physician assessment and guideline-based diagnostic criteria as the reference standard. AUC will be reported with 95% confidence intervals.

SECONDARY OUTCOMES:
Diagnostic performance of the AI model in clinically relevant subgroups. | At the nearest Heart Team meeting following the echocardiographic examination (typically within 1 week).
  Diagnostic performance of the AI model (AUC, sensitivity, specificity) in clinically relevant subgroups, such as patients with atrial fibrillation or subtypes of low-gradient aortic stenosis (classic, paradoxical, normal flow).

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Hryniewiecki, Professor of Medicine, Study Chair — Department of Valvular Heart Disease, National Institute of Cardiology, Warsaw, Poland; Michał Wrzosek, MD, Principal Investigator — Department of Valvular Heart Disease, National Institute of Cardiology, Warsaw, Poland; Karina Zatorska, MD, PhD, Study Director — Department of Valvular Heart Disease, National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Department of Valvular Heart Disease, National Institute of Cardiology, Warsaw, Poland, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wrzosek M, Buchwald M, Czernik P, Kupinski S, Zatorska K, Jasinska A, Zakrzewski D, Pukacki J, Mazurek C, Pekal R, Hryniewiecki T. Diagnosing Severe Low-Gradient vs Moderate Aortic Stenosis with Artificial Intelligence Based on Echocardiography Images. J Imaging Inform Med. 2025 Apr 21. doi: 10.1007/s10278-025-01497-4. Online ahead of print. PMID 40259202